CLINICAL TRIAL: NCT01673009
Title: Phase II Study of Gleevec/Imatinib Mesylate (STI-571, NCS 716051) in Neurofibromatosis (NF1) Patients With Plexiform Neurofibromas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0512-25
Record Dates: First submitted 2012-08-22; First posted 2012-08-27 (Estimated); Results first posted 2016-04-06 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Neurofibromatosis
Keywords: Gleevec
MeSH Terms: conditions — Neurofibromatoses | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Administration of Gleevec (Experimental): Gleevec® will be dosed orally 440 mg/m^2/day (max 800 mg/day) for pediatric subjects and 800 mg/day for adult patients.
  Interventions: Drug: Gleevec

INTERVENTIONS:
Drug: Gleevec — Gleevec® will be dosed orally 440 mg/m^2/day (max 800 mg/day) for pediatric subjects and 800 mg/day for adult patients.

SUMMARY:
THe primary objective is to estimate the response rate at 6 months to Gleevec® in patients with plexiform neurofibromas

DETAILED DESCRIPTION:
This is an open-label Phase II Study to determine the efficacy of Gleevec® in neurofibromatosis (NF1) patients with plexiform neurofibromas with the secondary goals of determining the toxicity, and tumor markers in this genetically defined population. The rationale for this study arises from the response of human and murine NF1 cells to Gleevec® in vitro and the response of a single NF1 patient treated with Gleevec® for airway compression by a plexiform neurofibroma with a dramatic response not previously seen in NF1 therapy. The plan of therapy will include oral dosing of Gleevec® at 440 mg/m^2/day (max 800 mg/day) for pediatric subjects and 800 mg/day for adult patients. (with 25% dose reduction for significant toxicity). Treatment will continue for 6 months with an option to continue as long as the patient remains on study provided the patient shows benefit from treatments with Gleevec® and there are no safety concerns.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 3-65 years of age.
2. Diagnosis of neurofibromatosis (NF1), as outpatients.
3. Presence of clinically significant plexiform neurofibromas (biopsy proven if possible with tissue blocks available); that is tumors that are potentially life threatening or are impinging on vital structures or significantly impair the quality of life from pain or other symptoms.
4. Patients must have measurable disease by magnetic resonance imaging (MRI). Patients must have a Karnofsky or Lansky Performance score of > 80% and a life expectancy of > 2 months.
5. Adequate end organ function, defined as the following:

   total bilirubin < 1.5 x ULN, SGOT and SGPT < 2.5 x UNL, creatinine < 1.5 x ULN, ANC > 1.5 x 109/L, platelets > 100 x 109/L.
6. Female patients of childbearing potential must have negative pregnancy test within 7 days before initiation of study drug dosing. Postmenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential. Male and female patients of reproductive potential must agree to employ an effective barrier method of birth control throughout the study and for up to 3 months following discontinuation of study drug.
7. Written, voluntary informed consent.

Exclusion criteria:

1. Patient has received any other investigational agents within 28 days of first day of study drug dosing, unless the disease is rapidly progressing.
2. Patient is < 5 years free of another primary malignancy except: if the other primary malignancy is not currently clinically significant nor requiring active intervention, or if other primary malignancy is a basal cell skin cancer or a cervical carcinoma in situ. Existence of any other malignant disease is not allowed.
3. Patient with Grade III/IV cardiac problems as defined by the New York Heart Association Criteria. (i.e., congestive heart failure, myocardial infarction within 6 months of study)
4. Female patients who are pregnant or breast-feeding.
5. Patient has a severe and/or uncontrolled medical disease (i.e., uncontrolled diabetes, chronic renal disease, or active uncontrolled infection).
6. Patient has a known brain metastasis. Non-specific CNS changes on MRI/CT characteristic of NF1 are allowed, but not known CNS malignancies.
7. Patient has known chronic liver disease (i.e., chronic active hepatitis, and cirrhosis).
8. Patient has a known diagnosis of human immunodeficiency virus (HIV) infection.
9. Patient received chemotherapy within 4 weeks (6 weeks for nitrosourea or mitomycin-C) prior to study entry, unless the disease is rapidly progressing.
10. Patient previously received radiotherapy to greater than 25 % of the bone marrow
11. Patient had a major surgery within 2 weeks prior to study entry.
12. Patient with any significant history of non-compliance to medical regimens or with inability to grant reliable informed consent.

Ages: 3 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2006-05; Primary Completion 2011-12 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Robertson KA, Nalepa G, Yang FC, Bowers DC, Ho CY, Hutchins GD, Croop JM, Vik TA, Denne SC, Parada LF, Hingtgen CM, Walsh LE, Yu M, Pradhan KR, Edwards-Brown MK, Cohen MD, Fletcher JW, Travers JB, Staser KW, Lee MW, Sherman MR, Davis CJ, Miller LC, Ingram DA, Clapp DW. Imatinib mesylate for plexiform neurofibromas in patients with neurofibromatosis type 1: a phase 2 trial. Lancet Oncol. 2012 Dec;13(12):1218-24. doi: 10.1016/S1470-2045(12)70414-X. Epub 2012 Oct 23. PMID 23099009

RESULTS

PARTICIPANT FLOW:
Groups:
- Administration of Gleevec: Gleevec® will be dosed orally 440 mg/m2/day (max 800 mg/day) for pediatric subjects and 800 mg/day for adult patients.
  Gleevec: Gleevec® will be dosed orally 440 mg/m2/day (max 800 mg/day) for pediatric subjects and 800 mg/day for adult patients.
Period: Overall Study
Arm/Group | Administration of Gleevec
Started | 36
Completed | 23
Not Completed | 13
Not completed — Physician Decision | 5
Not completed — Withdrawal by Subject | 8

BASELINE CHARACTERISTICS:
Arm/Group | Administration of Gleevec
Number analyzed (Participants) | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 25
  Between 18 and 65 years | 11
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 34
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 32
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Tumor Volume at 6 Months
Description: Volumetric measures were performed using MRI scan analysis. Response criteria include greater than 20 percent decrease in tumor volume as responsive. Greater than 20 percent increase in tumor volume as tumor progression. Less then 20 percent increase or decrease in tumor volume is stable disease
Time Frame: baseline to 6 months
Measure: Median (95% Confidence Interval); unit: percentage change of tumor volume
Arm/Group | Administration of Gleevec
Number analyzed (Participants) | 23
percentage change of tumor volume | 17 [6 to 33]

2. Secondary Outcome: Serum Bioactivity
Description: The investigators will quantitate the biologic activity of patient serum on fibroblast proliferation, migration, and collagen synthesis pre and post-Gleevec (7 days and 1 month)
Time Frame: 7 days and 1 month
Population: unable to measure this outcome because assay became unavailable
Arm/Group | Administration of Gleevec
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Administration of Gleevec
Serious Adverse Events (participants affected / at risk) | 1/36
Other Adverse Events (participants affected / at risk) | 12/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Administration of Gleevec (N=36)
liver dysfunction/failure (Hepatobiliary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Administration of Gleevec (N=36)
Rash (Skin and subcutaneous tissue disorders) | 4 (5)
Edema (General disorders) | 3 (4)
Pain (Nervous system disorders) | 3 (4)
Neutropenia (Investigations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes